CLINICAL TRIAL: NCT00423306
Title: A Phase-II Trial of ZIO 101 in Advanced Hepatocellular Carcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Alaunos Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SGL2005
Record Dates: First submitted 2007-01-16; First posted 2007-01-18 (Estimated); Last update posted 2013-11-14 (Estimated); Status verified 2013-11

CONDITIONS: HEPATOCELLULAR CARCINOMA
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — darinaparsin

ARMS (1):
- Single Arm (Experimental)
  Interventions: Drug: Darinaparsin

INTERVENTIONS:
Drug: Darinaparsin — 420 mg/m2 of Darinaparsin given twice weekly for three weeks, followed by one week of rest, for up to 6 months
  Other Names: ZIO-101

SUMMARY:
The study of safety of a new organic arsenic compound in the treatment of advanced hepatocellular carcinoma

ELIGIBILITY:
Inclusion Criteria

1. HCC diagnosed by histology or clinical evidence supported by liver mass(es) at least 2cm in the longest diameter and AFP equal to or more than 500 ng/mL in cirrhosis or chronic HBV or HCV infection27.
2. Male or female patients ≥ 18 years of age
3. Patients who have a life expectancy of at least 12 weeks
4. Patients who have at least one uni-dimensional measurable lesion by CT-scan or MRI according to Response Evaluation Criteria in Solid Tumors (RECIST).
5. Patients who have an Eastern Co-operative Oncology Group (ECOG) performance status of 0 - 2 (see Appendix 4).
6. Patients who have received local therapy, such as surgery, radiation therapy, hepatic arterial embolization, chemo-embolization, radio-frequency ablation or cryo-ablation are eligible, provided that they either have a target lesion which has not been subjected to local therapy and/or the target lesion(s) within the field of the local therapy has shown an increase of ≥ 25% in the size. Furthermore, the local therapy applied to target or non-target lesions needs to have been completed at least 8 weeks prior to study inclusion. Lesions treated with external beam radiation therapy are not acceptable as target lesions, unless they fulfil the conditions described above.
7. No more than one prior chemotherapy based regimen is allowed. Patients can receive up to two regimes where target therapies have been used (washout)
8. Cirrhotic status of Child-Pugh Class A or B only (Appendix 5).
9. Adequate hepatic function at screening as assessed by the following:

   * Platelet count ≥ 60 x 109/L
   * Hemoglobin ≥ 8.5 g/dl
   * Total bilirubin ≤ 3 mg/dl
   * ALT and AST ≤ 5 x upper limit of normal
   * Serum creatinine ≤ 2.0 x the upper limit of normal
   * PT-INR ≤ 2.3 or PT ≤ 6 seconds above control
10. Patients who give written informed consent prior to any study specific screening procedures with the understanding that the patient has the right to withdraw from the study at any time, without prejudice.

Exclusion Criteria

1. Previous malignancy (except for cervical carcinoma in situ, adequately treated basal cell carcinoma, or superficial bladder tumors [Ta, Tis and T1] or other malignancies curatively treated > 2 years prior to entry)
2. Congestive heart failure > NYHA Class II
3. Cardiac arrhythmias requiring anti-arrythmics (excluding beta blockers or digoxin for chronic stable atrial fibrillation) or QTc greater than 450 msec.
4. Active coronary artery disease or cardiac ischemia
5. Active clinically serious bacterial, viral or fungal infections (> grade 2 NCI-CTCAE, Version 3)
6. Known history of human immunodeficiency virus (HIV) infection for less than 2 years or uncontrolled disease on antiretroviral medication
7. Metastatic brain or meningeal tumors
8. Patients with seizure disorder requiring medication (such as anti-epileptics)
9. History of confusion or dementia or neurological condition that could mask a potential adverse response to the study drug (or something along these lines)
10. History of organ allograft
11. Substance abuse, medical, psychological or social conditions that may interfere with the patient's participation in the study or evaluation of the study results
12. Known or suspected allergy to the investigational agent or any agent given in association with this trial
13. Any condition that is unstable or which could jeopardize the safety of the patient and his/her compliance in the study
14. Pregnant or breast-feeding patients. Women of childbearing potential must have a negative pregnancy test performed within 14 days prior to the start of study drug. Both men and women enrolled in this trial must use adequate barrier birth control measures during the course of the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2007-01; Primary Completion 2013-12 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Response Rate | 6 months

SECONDARY OUTCOMES:
Survival (overall and progression free) | 6 months
toxicities | 6 months

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Miami, Florida
  - Atlanta, Georgia
  - Boston, Massachusetts
  - Kansas City, Missouri
  - New York, New York
  - Seattle, Washington